CLINICAL TRIAL: NCT03990246
Title: Impact of Emulsion Droplet Physical Properties on Postprandial Lipemia and Satiety in Healthy Adult Males
Brief Title: Emulsion Lipid Digestion & Satiety Study - Effect of Physical State and Acid Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-04-003
Record Dates: First submitted 2019-06-12; First posted 2019-06-18 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acid stable emulsion with solid droplets (Experimental): Acid stable emulsion with solid droplets will be consumed by participants in one study visit along with 1500 mg of crushed and dissolved acetaminophen.
  Interventions: Other: Acid stable emulsion with solid droplets
- Acid stable emulsion with liquid droplets (Experimental): Acid stable emulsion with liquid droplets will be consumed by participants in one study visit along with 1500 mg of crushed and dissolved acetaminophen.
  Interventions: Other: Acid stable emulsion with liquid droplets
- Acid unstable emulsion with solid droplets (Experimental): Acid unstable emulsion with solid droplets will be consumed by participants in one study visit along with 1500 mg of crushed and dissolved acetaminophen.
  Interventions: Other: Acid unstable emulsion with solid droplets
- Acid unstable emulsion with liquid droplets (Experimental): Acid unstable emulsion with liquid droplets will be consumed by participants in one study visit along with 1500 mg of crushed and dissolved acetaminophen.
  Interventions: Other: Acid unstable emulsion with liquid droplets

INTERVENTIONS:
Other: Acid stable emulsion with solid droplets — This will be a 250 mL acid stable beverage emulsion in which the droplets are crystalline. It will have identical similar to the other intervention, i.e. in a set of samples the emulsion lipid droplets are in the liquid state and are either acid stable or unstable and, in the other set of samples they are solid (i.e. crystallized) and are also either acid stable or unstable in the acidic environment of the stomach, and will be introduced at least 7 days apart. The emulsion will contain 20% of the lipid palm stearin with 2.2% of the emulsifier sorbitan monooleate (Tween80)
  Arms: Acid stable emulsion with solid droplets
Other: Acid stable emulsion with liquid droplets — This will be a 250 mL acid stable beverage emulsion in which the droplets are liquid. It will have identical similar to the other intervention, i.e. in a set of samples the emulsion lipid droplets are in the liquid state and are either acid stable or unstable and, in the other set of samples they are solid (i.e. crystallized) and are also either acid stable or unstable in the acidic environment of the stomach, and will be introduced at least 7 days apart. The emulsion will contain 20 % of the lipid palm olein with 2.2% of the emulsifier sorbitan monooleate (Tween80)
  Arms: Acid stable emulsion with liquid droplets
Other: Acid unstable emulsion with solid droplets — This will be a 250 mL acid unstable beverage emulsion in which the droplets are solid. It will have identical similar to the other intervention, i.e. in a set of samples the emulsion lipid droplets are in the liquid state and are either acid stable or unstable and, in the other set of samples they are solid (i.e. crystallized) and are also either acid stable or unstable in the acidic environment of the stomach, and will be introduced at least 7 days apart. The emulsion will contain 20% of the lipid palm stearin with 2.5% of the emulsifier sorbitan monostearate (Span60)
  Arms: Acid unstable emulsion with solid droplets
Other: Acid unstable emulsion with liquid droplets — This will be a 250 mL acid unstable beverage emulsion in which the droplets are liquid. It will have identical similar to the other intervention, i.e. in a set of samples the emulsion lipid droplets are in the liquid state and are either acid stable or unstable and, in the other set of samples they are solid (i.e. crystallized) and are also either acid stable or unstable in the acidic environment of the stomach, and will be introduced at least 7 days apart. The emulsion will contain 20 % of the lipid palm olein with 2.5% of the emulsifier sorbitan monostearate (Span60)
  Arms: Acid unstable emulsion with liquid droplets

SUMMARY:
The purpose of this study is to compare the changes in blood lipids and feelings of satiety after consumption of acid stable or acid unstable oil-in-water emulsions in which the droplets are in either the liquid or partially solid (i.e. crystalline) states.

DETAILED DESCRIPTION:
A double blinded randomized cross-over acute meal study will be carried out in which 15 healthy male participants will attend four study visits, separated by at least one week. On each study visit, fasted participants will consume either the emulsion with solid or liquid droplets and that is either acid stable or acid unstable, in a randomized order. All emulsions will have similar compositions, mainly differing in terms of droplet physical state, achieved by using lipids with different melting temperature. The emulsions will also contrast in terms of colloidal stability to acids, achieved by using different emulsifiers. This will isolate the impacts of physical state and acid stability, and their interactions. Postprandial lipemia, gastric emptying and satiety will be measured for 6 hours after consumption of each test beverage. The study meals will include crushed acetaminophen, the appearance of which will be measured in plasma as a measure of liquid content gastric emptying. It will also include periodic measurements of the gastric antrum area by ultrasound to assess the rate of gastric emptying. Participants will be asked to maintain their usual lifestyle habits throughout the study, with some changes in the 48 hour period leading up to each of the four visits.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18 - 26 kg/m2
* generally healthy
* non-smoking
* non to moderate alcohol drinkers
* fasting plasma cholesterol level <5.2 mmol/L
* plasma triacylglycerol level <1.7 mmol/L
* plasma glucose level <5.6 mmol/L
* no history of gastric surgeries

Exclusion Criteria:

* History of major medical conditions
* taking prescription medications/ over the counter medications
* taking natural health products/ dietary supplements (other than a multivitamin)
* oral antibiotic use in the previous 3 months
* planning to take oral antibiotics in the next 3 months
* food allergy/anaphylactic/life-threatening allergy
* smokers/ regular users of recreational drugs
* elite/ training athletes
* significant weight loss/ gain during the past 3 months
* previous reaction/ sensitivity to acetaminophen
* inability to avoid taking acetaminophen for 48 hours
* sensitivity to the artificial sweetener Sugar Twin® Sucralose and artificial vanilla extract
* not willing to consume Sugar Twin® Sucralose or Artificial vanilla.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in triacylglycerol blood concentrations | 6 hours
  Based on determination of fasting and postprandial blood triacylglycerol concentration (mmol/L)

SECONDARY OUTCOMES:
Participant visual analogue scale ratings of feelings of satiety | 6 hours
  Visual analogue scale ratings of feelings of hunger, fullness, appetite, prospective food consumption, desire to eat, and nausea after consuming the emulsion beverage. 0: not hungry, empty, no appetite, very little food, no desire to eat and no nausea, and 10: very hungry, very full, high appetite, a lot of food, very strong desire to eat and very nauseated. The distance from the left end of the scale will be measured (cm)
Rate of gastric emptying by measuring the changes in acetaminophen blood concentrations | 6 hours
  The rate of appearance of acetaminophen (consumed crushed in water immediately after test meal) in the plasma will be determined (mg/L)
Changes in fatty acid concentration of blood triacylglycerols | 6 hour
  Analysis based on fasting and postprandial blood sample analysis (mmol/L)
Changes in satiety hormone blood concentrations | 6 hours
  Analysis of blood for Ghrelin, Leptin, GLP-1,PYY, GIP, and Insulin, at fasting and postprandially (pg/mL)
Changes in concentrations of inflammatory blood markers (ug/mL) | 6 hours
  Analysis of blood for CD14 and LBP at fasting and postprandially
Rate of gastric emptying by measuring the change in the gastric antrum area | 6 hours
  Determined by measuring the cross-sectional area of the gastric antrum using ultrasound (cm*cm)
Changes in glucose blood concentrations | 6 hour
  Based on determination of fasting and postprandial blood glucose (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Hamad S, Tari NR, Mathiyalagan G, Wright AJ. Emulsion acid colloidal stability and droplet crystallinity modulate postprandial gastric emptying and short-term satiety: a randomized, double-blinded, crossover, controlled trial in healthy adult males. Am J Clin Nutr. 2021 Sep 1;114(3):997-1011. doi: 10.1093/ajcn/nqab116. PMID 33963742
- [Derived] Hamad S, Thilakarathna SH, Cuncins A, Brown M, Wright AJ. Emulsion Droplet Crystallinity Attenuates Short-Term Satiety in Healthy Adult Males: A Randomized, Double-Blinded, Crossover, Acute Meal Study. J Nutr. 2020 Sep 1;150(9):2295-2304. doi: 10.1093/jn/nxaa164. PMID 32556204